CLINICAL TRIAL: NCT05494164
Title: Effect of Nigella Sativa on Selected Outcomes Among Patients With Chronic Rhinosinusitis: Prospective Clinical Trial
Brief Title: Nigella Sativa for Selected Outcomes in Chronic Rhinosinusitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reham Samir Fatehallah, Assistant Lecturer at Medical-Surgical Nursing, Faculty of Nursing, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-03
Record Dates: First submitted 2022-08-05; First posted 2022-08-09 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Chronic Rhinosinusitis
Keywords: Nigella sativa; chronic rhinosinusitis; nasal oil drops; outcomes

STUDY DESIGN:
Who Masked: Participant
Masking Description: participants in both groups will be blinded to which treatment arms they will be assigned to till the end of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Nigella sativa nasal oil drops
  Interventions: Other: Nigella sativa nasal oil drops; Drug: standard treatment
- Control group (Other): standard treatment
  Interventions: Drug: standard treatment

INTERVENTIONS:
Other: Nigella sativa nasal oil drops — in addition to the standard treatment, the study group will receive one nasal drop of the prepared N. sativa nasal oil drops in each nostril twice daily which are equivalent to a daily dose of 100 milligram of a pure N. sativa oil for four weeks. N. sativa oil was prepared from N. sativa seeds and it was mixed in Sesame oil with a ratio of 1 to 1. The prepared drops will then be placed in dark containers with a specific dropper. Each participant will be instructed regarding the dose, proper position and steps, assisted by a flyer which will be developed by the researcher.
  Arms: Study group
Drug: standard treatment — intranasal corticosteroids in addition to nasal irrigation with sea water; for patients with allergy the standard treatment is oral antihistamines with or without oral corticosteroids.

SUMMARY:
the study is intended to test the effect of Nigella sativa nasal oil drops on selected outcomes among patients with chronic rhinosinusitis using prospective clinical trial design. To achieve the aim of the current trial the following research hypotheses are postulated: H1. The total severity of symptoms mean scores of patients with CRS who will use Nigella sativa nasal oil drops will be different from the total severity of symptoms mean scores of a control group.

H2. The total sleep quality mean scores of patients with CRS who will use Nigella sativa nasal oil drops will be different from the total sleep quality mean scores of a control group.

H3. The total patient satisfaction mean scores of patients with CRS who will use Nigella sativa nasal oil drops will be different from the total patient satisfaction mean scores of a control group.

DETAILED DESCRIPTION:
The clinical trial will be conducted to examine the effect of administering a daily dose of 100 mg Nigella sativa nasal oil drops for four weeks on selected outcomes which include severity of symptoms, sleep quality and patient satisfaction among patients with chronic rhinosinusitis. The trial will be conducted on 102 adult patients with chronic rhinosinusitis who will be randomly assigned to either a study group (51 participant) who will receive Nigella sativa beside the standard treatment or a control group (51 participant) who will receive the standard treatment only. The current trial will be conducted in the Ear, Nose and Throat (ENT) outpatient clinic at Kasr Al Ainy University Hospital, Cairo, Egypt. Required data will be collected by using the following four tools: (a) Demographic and Medical Data Form (DMDF), (b) Sino-Nasal Outcome Test 22 (SNOT-22), (c) Sleep Quality Scale (SQS) and (d) Treatment Satisfaction Questionnaire for Medication (TSQM). The researcher prepared a flyer that will be handed in for the study group to explain how the oil will be utilized by the participants. The formal initial approval was obtained from Research Ethics Committee at Faculty of Nursing, Cairo University and an official permission was also obtained from the hospital administrators for conducting the trial. The researcher collaborated with Emeritus Professor in Pharmacognosy from the College of Pharmacy for the preparation of N. sativa nasal oil drops from Nigella sativa and Sesame seeds. Thereafter, data collection will be carried out from both groups using the following five steps as follows: recruitment and randomization; interviewing; initial assessment; intervention; follow-up and monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients from 18 to 60 years old,
* able to communicate,
* having a confirmed diagnosis of CRS by signs and symptoms and meeting the criteria of having twelve consecutive weeks or longer of two or more of the following signs and symptoms will be recruited for the current trial: (a) mucopurulent drainage, (b) nasal obstruction/congestion, (c) facial pain-pressure-fullness and (d) decreased sense of smell; and one or more of the following signs and symptoms: (a) purulent mucus or edema in middle meatus or anterior ethmoid region or (b) radiographic imaging showing sinus inflammation.

Exclusion Criteria:

* Pregnancy,
* lactating mothers,
* immunodeficiency,
* scheduled for surgical management for nasal polyposis,
* fever more than 37.8 ﹾC,
* patients with coagulation disorders or using anticoagulants,
* patients taking non-potassium sparing diuretics,
* patients allergic to N. sativa (patients reactive to sensitivity test)
* patients using any type of natural products as a complementary therapy at the time of the trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2022-08-07 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Severity of physiological symptoms as measured by Sino-Nasal Outcome Test 22 (SNOT-22) | from two to four weeks
  SNOT-22 consists of 22 items that measure four domains as follows: (a) nasal symptoms domain that contains eight items, (b) otologic symptoms domain which includes four items, (c) sleep symptoms domain which includes seven items and (d) emotional symptoms domain that contains three items. SNOT-22 is scored using a Likert scale where 0="No problem", 1="Very mild problem", 2="Mild or slight problem", 3="Moderate problem", 4="Severe problem" and 5="Problem as bad as it can be". The overall scores of the SNOT-22 is ranged from 0 to 110 with higher scores suggesting symptom severity.
Sleep quality as measured by Sleep Quality Scale (SQS) | from two to four weeks
  Sleep Quality Scale (SQS) consists of 28 items, which evaluate six domains of sleep quality as follows: (a) daytime dysfunction/symptoms which contain twelve items, (b) restoration after sleep which include four items, (c) difficulty falling asleep that contain four items, (d) difficulty getting up that include three items, (e) difficulty in maintaining asleep which contain two items and (f) satisfaction with sleep which include three items. Sleep Quality Scale is scored through a four-point, Likert-type scale; (0 = "few," 1 = "sometimes," 2 = "often," and 3 = "almost always"). Scores on items belong to factors 2 and 5 (restoration after sleep and satisfaction with sleep) are reversely scored. Total scores are ranged from 0 to 84, with higher scores denoting more acute sleep problems.

SECONDARY OUTCOMES:
severity of sleep and emotional symptoms as measured by Sino-Nasal Outcome Test 22 (SNOT-22) (sleep and emotional symptoms domains) | from two to eight weeks
  SNOT-22 consists of 22 items that measure four domains as follows: (a) nasal symptoms domain that contains eight items, (b) otologic symptoms domain which includes four items, (c) sleep symptoms domain which includes seven items and (d) emotional symptoms domain that contains three items. SNOT-22 is scored using a Likert scale where 0="No problem", 1="Very mild problem", 2="Mild or slight problem", 3="Moderate problem", 4="Severe problem" and 5="Problem as bad as it can be". The overall scores of the SNOT-22 is ranged from 0 to 110 with higher scores suggesting symptom severity.
patient satisfaction as measured by Treatment Satisfaction Questionnaire with Medications (TSQM) | from two to eight weeks
  Treatment Satisfaction Questionnaire for Medication includes 14 items that assess four key dimensions of treatment satisfaction: (a) effectiveness which includes three items, (b) side Effects which contain five items, (c) convenience that include three items and (d) global Satisfaction that contain three items. Item of TAQM are scaled on 5 or 7 point Likert scale, except one item which is answered with 1= "Yes" or 0= "No". Scores for each domain are calculated independently by adding the TSQM items in each domain and then transforming the composite score into a value ranging from 0 to 100; higher values indicate higher satisfaction, better perceived effectiveness, lower burden associated to side-effects, better convenience.

CONTACTS AND LOCATIONS:
Overall Officials: Reham S. Fatehallah, Master, Principal Investigator — Cairo University; Bassamat O. Ahmed, Doctorate, Study Director — Cairo University; Hanan A. Al Sebaee, Doctorate, Study Director — Cairo University; Fathy M. Soliman, Doctorate, Study Director — Cairo University; Adel El-Antably, Doctorate, Study Director — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No